CLINICAL TRIAL: NCT01332214
Title: A Randomised, Single-blind, Placebo-controlled Single-centre Phase I Study in Healthy Male Volunteers to Assess the Safety, Tolerability and Pharmacokinetics of AZD2820 After Single Ascending Doses
Brief Title: To Assess the Safety, Tolerability and Pharmacokinetics of AZD2820 After Single Ascending Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D3870C00001
Record Dates: First submitted 2011-04-06; First posted 2011-04-11 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Phase 1; healthy male volunteers; dose escalation; pharmacokinetics; Single Ascending Dose; AZD2820 Cmax; tmax; t1/2λz

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD2820 (Experimental)
  Interventions: Drug: AZD2820
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2820 — Subcutaneous Injection in abdomen or Thigh
  Arms: AZD2820
Drug: Placebo — Subcutaneous Injection in abdomen or Thigh
  Arms: Placebo

SUMMARY:
This is a randomised, single-blind, placebo-controlled Phase I study to investigate the safety, tolerability and pharmacokinetics after administration of single doses of AZD2820 to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male subjects aged ≥20 - ≤45 years with suitable veins for cannulation or repeated venepuncture.
* Male subjects should be willing to use barrier contraception ie, condoms, from the day of dosing until 3 months after dosing with the investigational product.
* Have a body mass index (BMI) between≥ 18 and ≤30 kg/m2 and weigh at least 50 kg and no more than 100 kg.
* Provision of signed, written and dated informed consent for genetic research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this Clinical Study Protocol, so long as they consent.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* A history of erectile dysfunction or anatomic abnormality of the penis (eg, cavernosal fibrosis, Peyronie's disease, or plaques) which interferes with normal erectile function
* Predisposition or history of priapism (eg, sickle cell anemia or trait).
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety variables ( Adverse events, Vital signs, ECG, EEG, Regiscan, Safety labs.) | Assessments performed multilpe times from the morning day 1 before dose until day 3. And then once at the follow up after 14-18 days

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of AZD2820 and assess the dose proportionality of the pharmacokinetics following single ascending doses of AZD2820 by assessment Cmax, tmax, t1/2 , AUC, CL/F, Ae and CLR. | Blood samples will be taken multiple times from the morning day 1 before dose until day 2

CONTACTS AND LOCATIONS:
Overall Officials: Mirjana Kujacic, PhD, Study Chair — AstraZeneca; Prof J Ritter BM BCh, MRCP, FRCP, Principal Investigator — Quintiles, Inc.; Mark Berner Hansen, PhD, Study Director — AstraZeneca
Locations (1):
- Research Site, London, United Kingdom